CLINICAL TRIAL: NCT00013221
Title: Exercise Effect on Aerobic Capacity and QOL in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NRI 95-213
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
Chronic heart failure (HF) is a syndrome of impaired ventricular function resulting in clinical symptoms of fatigue, dyspnea, and decreased exercise capacity. These symptoms lead to a cyclical pattern of an increasing sedentary lifestyle with accompanying deconditioning and deterioration of muscle function. Until recently, the prescription for individuals with HF was rest and minimization of physical exertion.

DETAILED DESCRIPTION:
Background:

Chronic heart failure (HF) is a syndrome of impaired ventricular function resulting in clinical symptoms of fatigue, dyspnea, and decreased exercise capacity. These symptoms lead to a cyclical pattern of an increasing sedentary lifestyle with accompanying deconditioning and deterioration of muscle function. Until recently, the prescription for individuals with HF was rest and minimization of physical exertion.

Objectives:

The primary objectives of this randomized clinical trial were to determine whether subjects, with moderate to severe chronic HF, who completed a 12-week individualized program of cardiopulmonary training (exercise group) would have significantly greater (i) quality of life, measured by the Rand Short Form-36, and (ii) aerobic fitness, measured by oxygen uptake during symptom limited maximal metabolic treadmill testing, than subjects who met weekly with an investigator and received vital sign measurements (non-exercise group).

Methods:

A randomized controlled clinical trial was utilized. Individuals who met the inclusion criteria were randomly assigned to either an exercise or control group. Individuals in the exercise group received 36 weeks of exercise training (primary outcome variables were measured at 12 weeks). Participants in the control group received weekly visits with a nurse for 12 weeks.

Status:

Ongoing data analysis for publication. Final report submitted.

ELIGIBILITY:
Inclusion Criteria:

Left ventricular ejection fraction less than or equal to 40%. Stable heart failure.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen G. Collins, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL; Walter Edwin Langbein, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

REFERENCES:
- [Result] Collins E, Langbein WE, Dilan-Koetje J, Bammert C, Hanson K, Reda D, Edwards L. Effects of exercise training on aerobic capacity and quality of life in individuals with heart failure. Heart Lung. 2004 May-Jun;33(3):154-61. doi: 10.1016/j.hrtlng.2003.12.009. PMID 15136775